CLINICAL TRIAL: NCT00891748
Title: A Phase I/IIa Study of Dose-escalating Intravesical AdCD40L Instillation in Urinary Bladder Carcinoma
Brief Title: Safety Study on AdCD40L Gene Therapy for Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Thomas H Totterman, Uppsala University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001:CD40L; 2006-000985-34
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2009-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AdCD40L (Experimental): Adenovirus vector serotype 5, E1/E3 deletion with human CD40L gene driven by RSV promoter.
  Interventions: Genetic: AdCD40L

INTERVENTIONS:
Genetic: AdCD40L — Adenovirus vector serotype 5, E1/E3 deletion with human CD40L gene driven by RSV promoter

SUMMARY:
The study objective is to evaluate the feasibility of three instillations of immunostimulating gene therapy (AdCD40L) in patients with urinary bladder cancer. Tolerance, toxicity and immunological parameters will be evaluated during and post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of transitional cell carcinoma of the bladder
* ECOG 0-2
* 18 years of age or older
* signed informed consent
* for the Phase I part: patient scheduled for cystectomy

Exclusion Criteria:

* Woman of childbearing potential (fertile woman)
* Other malignancy within 5 years of study, except for non-melanoma skin cancer
* Metastatic disease
* Previous exposure to any intravesical therapy for bladder cancer: within 3 months for chemotherapy and within 6 months for BCG therapy.
* Previous pelvic radiation or treatment with any cytotoxic, immunologic or chemotherapeutic agent for non-malignant conditions within 5 years of study.
* Clinically abnormal hepatic, renal or bone marrow function, or coagulation disorders in the opinion of the investigator.
* Chronic urinary tract infections.
* Serous infection of G.U. surgery, except for bladder cancer, within 1 month of study requiring more than 3 days of hospital care.
* Vesical capacity <150mL and/or vesical obstruction with residual >150 mL after spontaneous voiding.
* Previous exposure to any experimental drug within 3 months from enrolment.
* Any significant medical or psychiatric illness that would prevent the patient from giving informed consent of from following the study procedures.
* Patients who presently have urothelial cell carcinoma of the upper G.U. tract
* Patients with systemic autoimmune disease
* Patients that do not consent to that tissue and blood samples are stored in a biobank
* Treatment with systemically administered corticosteroids and NSAID within 4 weeks prior to first study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Toxicity | Continously during therapy and at follow up 30d

SECONDARY OUTCOMES:
Inflammation | Continously during treatment and at follow up 30d

CONTACTS AND LOCATIONS:
Overall Officials: Per-Uno Malmstrom, MD PhD, Principal Investigator — Uppsala University Hospital, Uppsala, Sweden
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden